CLINICAL TRIAL: NCT03709810
Title: A Randomized, Single-Blind, Clinical Study to Assess Food Occlusion Efficacy of a Marketed Denture Adhesive in Healthy, Edentulous Subjects
Brief Title: A Study to Investigate Food Occlusion Efficacy of a Denture Adhesive in Denture Wearers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 209649
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Denture Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Test Denture Adhesive (Experimental): Test denture adhesive will be applied directly from the tubes using a continuous strip pattern to the upper and lower denture which will then be placed in mouth of the participants.
  Interventions: Combination Product: Marketed Denture Adhesive (Super Poligrip Max Seal)
- Control (Other): Participants will not apply any denture adhesive in this treatment arm.
  Interventions: Other: No Adhesive

INTERVENTIONS:
Combination Product: Marketed Denture Adhesive (Super Poligrip Max Seal) — The denture adhesive will be applied directly from the tubes. 1.6 g of adhesive per treatment will be applied to each participant's dentures. This dose will be split as 1.00±0.1 g for the maxillary and 0.6±0.1g for the mandibular dentures.
  Arms: Test Denture Adhesive
Other: No Adhesive — No adhesive will be applied.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the ability of a marketed denture adhesive to restrict food ingress underneath dentures during eating.

DETAILED DESCRIPTION:
This is a single center, controlled, single-blind, randomized, two-treatment, two-period, cross-over design in participants with full upper and lower dentures. The study hypothesis is that this methodology will enable comparisons between denture adhesives and no adhesive to demonstrate the effectiveness of denture adhesives in restricting food ingress under dentures during eating. This study will consist of three visits: Visit 1 - Screening Visit; Visit 2 - Treatment 1 Visit; Visit 3 - Treatment 2 Visit. Participants will use test product which is a marketed denture adhesive (Super Poligrip Max Seal [SPMS]) (application will be controlled by weight) to the dentures in a pattern of continuous strips which will be applied to upper and lower denture and will be then placed in mouth and participants will also use no adhesive as a control. Participants will cross-over between treatments so that all participants will participate in all 2 treatment arms. An hour after the participant has worn their denture, they will chew a portion of peanuts in a controlled manner. After a rinsing procedure with water, the dentures will be removed, and any peanuts that have been migrated under each denture will be collected and weighed after a drying process. Participants will also answer a short questionnaire on the procedure and record the number of times their denture dislodged during the chewing procedure. The number of denture dislodgments reported by the participants during the chewing of the peanuts will also be collected and analyzed and this, and the questionnaire data, will be used to support the findings of the peanuts mass measure.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is male or female who, at the time of screening, is between the ages of 18 and 85 years, inclusive.
* Participant who is willing and able to comply with scheduled visits, treatment plan and other study procedures.
* Participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant/relevant abnormalities in medical history or upon oral examination, or condition, that would impact the Participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Self-reports experience of getting food trapped under their denture.
* Is a habitual wearer of both of their dentures defined as participants who wear both of their dentures for the majority of their time whilst awake.
* Have denture protheses that fulfil all of the following: a) A qualifying conventional acrylic full denture in both the upper and lower arch; b) Dentures are well fitting (Kapur (Olshan Modification) Retention and Stability Index Sum Score ≥6) with no individual stability or retention scores <1; c) Dentures are well made (according to the well-made assessment); d) Has a peanut particle migration rating >0 for each denture.

Exclusion Criteria:

* A Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the Participant inappropriate for entry into this study.
* A Participant who is a pregnant female (self-reported).
* A Participant who is a breastfeeding female.
* A Participant with known or suspected intolerance or hypersensitivity to the study materials(or closely related compounds) or any of their stated ingredients.
* A Participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
* A Participant unwilling or unable to comply with the Lifestyle Considerations such as a) During the entire study Participants will not be permitted to have any dental/denture work performed during the time they are in the study, unless discussed and permitted by the examiner. This is to assure that the denture fit will not be altered during the study; b) During the treatment visits Participants will not be allowed to use tobacco or nicotine or nicotine-containing products following denture insertion until after their dentures are returned at completion of the food occlusion testing and Participants will not be allowed to use tobacco or nicotine or nicotine-containing products following denture insertion until after their dentures are returned at completion of the food occlusion testing.
* History of swallowing difficulties or choking.
* Currently taking or have taken a bisphosphonate drug (i.e., Fosamax, Actonel, Boniva).
* Any clinically significant or relevant oral abnormality (e.g. temporomandibular joint [TMJ] problems) that, in the opinion of the investigator, could affect the Participant's participation in the study.
* Known allergy to peanuts or any other nut.
* Any condition or medication which, in the opinion of the investigator, is currently causing xerostomia.
* Recent history (within the last year) of alcohol or other substance abuse.
* Oral soft tissue examination findings such as stomatitis, open sores, lesions, redness or swelling which in the opinion of the investigator, would interfere with the conduct of the study or the safety of the Participant.
* Use of any medication that, in the opinion of the investigator, would interfere with the conduct of the study.
* A serious chronic disease requiring intermittent hospital visits.
* Having been previously enrolled in this study.
* Any participant, in the opinion of the investigator, who should not participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=209649&attachmentIdentifier=c0b18f51-6094-46da-80ca-94161383820c&fileName=gsk-209649-protocol-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=209649&attachmentIdentifier=86b9402b-8782-44e2-a4d4-972bcf302724&fileName=gsk-209649-reporting-and-analysis-plan-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a single center in the United States. A total of 53 participants were screened, of which 49 were enrolled. 48 participants were randomized and completed the study.
Pre-assignment Details: Participants allocated to either intervention A(experimental test adhesive)or B(no adhesive)in period1. In period2,alternative sequence was assigned(B or A)in a crossover manner.Each period consisted of 1day testing(single use of experimental test product)with at least2days between adjacent treatment visits to recover from mastication procedures.
Groups:
- Sequence 1: Participants received interventions in a crossover manner: A (experimental denture adhesive) in period 1, then intervention B (no adhesive) in period 2.
- Sequence 2: Participants received interventions in a crossover manner: B (no adhesive) in period 1, then intervention A (experimental denture adhesive) in period 2.
Period: Treatment Period 1 (Visit 2)
Arm/Group | Sequence 1 | Sequence 2
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Treatment Period 2 (Visit 3)
Arm/Group | Sequence 1 | Sequence 2
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population (N=48) included all randomized participants who received at least 1 dose of the study product.
Groups:
- Overall: Included participants randomized in both the treatment arms
Arm/Group | Overall
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Food Occlusion Analysis of Combined Mass of Peanuts Under Combined Maxillary (Upper) and Mandibular (Lower) Dentures
Description: On each test day(Visit2,3)participants underwent an Oral Soft Tissue (OST) exam,dentures cleaned using denture cleanser.Product application controlled by weight:1g(+/-0.1g)to upper denture ,0.6g (+/-0.1g)to lower denture by dispensing staff. After60+/-5minutes(min) of replacing denture in the mouth,participants consumed 30-32g of non-salted peanuts, divided into smaller portions of approximately(app) 8nut halves. Each portion was chewed for app20 seconds(sec). After which mouth rinsed with water for app10sec. Both upper and lower dentures were removed,any nuts remaining in mouth were collected using gauze.Dentures and gauzes placed in beaker with warm de-ionized water and sonicated for 30min,water was strained by sieve.Collected nuts washed,air-dried and transferred to pre-weighed aluminium weighing pans,dried at 40-degree Celsius (deg C)for 5 hours(h). Pans removed,cooled to room temperature,weighed to determine mass of nuts collected from each denture.
Time Frame: Upto 16 days
Population: Efficacy analysis was performed on modified intent-to-treat (mITT) population [N=48] included all randomized participants who received at least 1 dose of the study product and had at least 1 on-therapy assessment of efficacy.
Measure: Geometric Mean (95% Confidence Interval); unit: Milligrams (mg)
Groups:
- Experimental Denture Adhesive: Participants randomized in this arm received 1.6 grams (g) of adhesive which was applied as 1.0 g (+/-0.1 g) on maxillary denture and 0.6 g (+/-0.1 g) on mandibular denture by dispensing staff. The adhesive was applied to upper and lower denture using a continuous strip pattern which was then placed in mouth for 60+/-5 min.
- No Adhesive: Participants did not receive any denture adhesive treatment randomized in this arm.
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 48 | 48
Milligrams (mg) | 5.56 [3.72 to 8.31] | 29.13 [19.48 to 43.56]
Statistical Analysis 1: Comparison: Experimental Denture Adhesive vs No Adhesive; Test type: Superiority; p < 0.0001, ANOVA; Log10 peanuts mass as response variable, study product and period as fixed explanatory effects, and participant as a random effect; Geometric Mean Ratio = 0.19, 95% CI 2-sided [0.12 to 0.30] — GMR=(Experimental denture adhesive/ No Adhesive)

2. Secondary Outcome: Food Occlusion Analysis of Mass of Peanuts Under Maxillary Denture
Description: On each test day (Visit2,3) participants underwent an OST exam, dentures cleaned using denture cleanser. Product application controlled by weight:1g(+/-0.1g)to upper denture ,0.6g (+/-0.1g)to lower denture by dispensing staff. After 60+/-5 min of replacing denture in the mouth, participants consumed 30-32g of non-salted peanuts, divided into smaller portions of app 8nut halves. Each portion was chewed for app20 sec. After which mouth rinsed with water for app10sec. Both upper and lower dentures were removed, any nuts remaining in mouth were collected using gauze. Dentures and gauzes placed in beaker with warm de-ionized water and sonicated for 30min, water was strained by sieve. Collected nuts washed, air-dried and transferred to pre-weighed aluminium weighing pans, dried at 40-deg C for 5h. Pans removed, cooled to room temperature, weighed to determine mass of nuts collected from each denture.
Time Frame: Upto 16 days
Population: Efficacy analysis was performed on mITT population [N=48] included all randomized participants who received at least 1 dose of the study product and had at least 1 on-therapy assessment of efficacy.
Measure: Geometric Mean (95% Confidence Interval); unit: mg
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 48 | 48
mg | 1.39 [0.92 to 2.11] | 8.17 [5.39 to 12.38]

3. Secondary Outcome: Food Occlusion Analysis of Mass of Peanuts Under Mandibular Denture
Description: as for outcome 2
Time Frame: Upto 16 days
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mg
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 48 | 48
mg | 2.75 [1.63 to 4.64] | 13.07 [7.75 to 22.02]

4. Secondary Outcome: Number of Denture Dislodgements During Chewing as Reported by Participants
Description: On each test day (Visit 2,3) participants had an OST exam and their dentures were cleaned before study product was applied to the dentures. 1g (+/-) was applied to the upper denture and 0.6g (+/-) was applied to the lower dentures by dispensing staff. After insertion of the dentures into participants mouths, they were required to wait 60 mins (+/- 5mins) after which they were required to chew 30-32g of non-salted peanuts, divided into smaller portions of approximately 8 nut halves. Participants were required to chew each portion of peanuts for approximately 20 secs. Whilst consuming the peanuts, participants were required to tick a box every time they felt their denture dislodge. The total number of dislodgments were recorded by study site staff.
Time Frame: Upto 16 days
Population: as for outcome 2
Measure: Median (Full Range); unit: Number of denture dislodgements
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 48 | 48
Number of denture dislodgements | 0.0 [0 to 10] | 4.0 [0 to 28]

5. Secondary Outcome: Mean Scores From Participant Completed Questionnaire
Description: On each test day(Visit 2,3)participants underwent an OST exam,dentures cleaned using denture cleanser. Product application controlled by weight:1g(+/-0.1g)to upper denture,0.6g (+/-0.1g)to lower denture by dispensing staff. After 60+/-5min of replacing denture in the mouth, participants consumed 30-32g of non-salted peanuts, divided into smaller portions of app8nut halves. Each portion chewed for app20 sec. After eating all,participants answered a questionnaire for chewing experience by questions (Q):Q1,were you aware of nuts pieces under your denture:yes/no.Participants answered no to Q1 were not required to answerQ2,3;they were automatically assigned 0 score for Q2,3. Participants who answered yes to Q1 were asked Q2,3;Q2,rate amount of nuts pieces under your denture on0-10scale;Q3,how bothered were you by nuts pieces went under your denture on0-10scale.Q2score:0=none,10=lots of nuts pieces;Q3score:0=not at all bothered,10=extremely bothered. Lower scores indicate better results.
Time Frame: Upto 16 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Experimental Denture Adhesive | No Adhesive
Number analyzed (Participants) | 48 | 48
Score on scale
  Amount of peanut pieces under denture | 0.8 (0.29) | 3.8 (0.52)
  Bothered by peanut pieces under denture | 0.7 (0.28) | 4.0 (0.57)

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form until 5 days after last administration of study drug (or last procedure)
Description: Safety population: all randomized participants who received at least one dose of study medication. All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious adverse events (SAEs) were collected and reported.
Arm/Group | Experimental Denture Adhesive | No Adhesive
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 2/48 | 4/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Denture Adhesive (N=48) | No Adhesive (N=48)
Oral hyperkeratosis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mouth Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue biting (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT03709810/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT03709810/SAP_001.pdf